CLINICAL TRIAL: NCT04116047
Title: Phase III Randomised Controlled Trial Comparing Alternative Regimens for Escalating Treatment of Intermediate and High-risk Oropharyngeal Cancer
Brief Title: CompARE: Escalating Treatment of Intermediate and High-risk Oropharyngeal Cancer (OPC)
Acronym: CompARE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: AstraZeneca (Industry); Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG 14-093; 2014-003389-26 (EudraCT Number); ISRCTN41478539 (Registry Identifier: International Standard Randomised Clinical Trial Number)
Record Dates: First submitted 2018-08-13; First posted 2019-10-04 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Oropharyngeal Cancer
Keywords: Oropharyngeal cancer; HPV
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Cisplatin; durvalumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (control): chemoradiotherapy (Active Comparator): Concomitant chemoradiotherapy, 3-weekly cisplatin 100mg/m2 or weekly 40mg/m2 with Intensity Modulated Radiotherapy (IMRT) using 70 gray (Gy) in 35F(fractions) +/- neck dissection as indicated by clinical and radiological assessment 3-months post treatment. This is the international gold standard.
  Interventions: Drug: Cisplatin; Procedure: Radiotherapy
- Arm 5: Durvalumab + Arm 1 (Experimental): One dose of induction durvalumab 1500mg by intravenous (IV) infusion followed by arm 1 within four weeks. Within one-two weeks after the completion of arm 1, durvalumab 1500mg every four weeks will be initiated for a total of 6 months
  Interventions: Drug: Cisplatin; Drug: Durvalumab; Procedure: Radiotherapy

INTERVENTIONS:
Drug: Cisplatin
  Other Names: CDDP, Platinol
Drug: Durvalumab
  Other Names: MEDI-4736, Imfinzi
  Arms: Arm 5: Durvalumab + Arm 1
Procedure: Radiotherapy

SUMMARY:
CompARE is a multicentre, phase III open-label randomised controlled trial using an adaptive, Multi-Arm, Multi-Stage (MAMS) design.

DETAILED DESCRIPTION:
The CompARE Trial examines alternative regimens for escalating treatment of intermediate and high-risk oropharyngeal cancer in an adult patient population. The aim is to assess whether escalated radiotherapy, adding surgery or immunotherapy will improve overall survival and quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Oropharyngeal squamous cell carcinoma (OPSCC) in base of tongue and tonsil with a Multidisciplinary Team (MDT) recommendation for treatment with definitive concurrent chemoradiotherapy
2. All OPC T4 or N3 (HPV+ and HPV-) OR all HPV -ve (negative) OPC T1-T4, N1-N3 or T3-4, N0 OR HPV +ve (positive) OPC T1-T4 with N2b-N3 nodes AND who are smokers ≥ 10 pack years current or previous smoking history
3. Minimum life expectancy of 3 months
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Adequate renal function, glomerular filtration rate (GFR) >50ml/min calculated using Cockcroft-Gault formula
6. Adequate bone marrow function (absolute neutrophil count (ANC) ≥1.5 x 109/L, haemoglobin ≥9.0g/dL and platelets ≥100 x 109/L)
7. Adequate liver function i.e. plasma bilirubin ≤1.5 times the upper limit of normal (ULN), and alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤2.5 x ULN
8. Prothrombin time (PT) ≤1.5 x ULN or International Normalised Ratio (INR) ≤1. 5
9. Magnesium ≥ lower limit of normal
10. No cancers in previous 5 years, except basal cell carcinoma of skin and cervical intra-epithelial neoplasia (CIN)
11. Aged 18-70
12. Written informed consent given for the trial
13. Surgically resectable disease if being randomised to all four arms
14. Females must either be of non-reproductive potential (i.e. post-menopausal by history: ≥55 years old and no menses for ≥1 year without an alternative medical cause; or history of hysterectomy, or history of bilateral tubal ligation or history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
15. Willingness to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. All T1-T2,N0 OPC (HPV +ve or HPV-ve)
2. HPV positive patients who are:

   T1-T3, N0-N2c non-smokers T1-T3, N0-N2c smokers with ≤10 pack years or T1-T2, N0-N2a smokers with ≥10 pack years
3. Unfit for chemoradiotherapy regimens
4. Creatinine Clearance <50ml/min
5. Treatment with any of the following, prior to randomisation:

   1. Any Investigational Medicinal Products (IMP) within 30 days
   2. Any other chemotherapy, immunotherapy or anticancer agents within 3 weeks
   3. Major surgery within 4 weeks
6. History of allergic reactions to any of the IMPs and excipients used in this trial
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C, Human Immunodeficiency Virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
8. Women who are pregnant or breast-feeding. Women of child- bearing potential must have a negative pregnancy test performed within 7 days prior to randomisation
9. Men or women who are not prepared to practise methods of contraception of proven efficacy during treatment and for 6 months following the end of treatment
10. Any condition that, in the opinion of the Investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

    Additional Exclusion Criteria for Arm 5 only:
11. Any previous treatment with PD-L or PD-L1 inhibitor, including durvalumab
12. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid dose
13. Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease e.g. colitis or Crohn's disease, diverticulitis (with the exception of diverticulosis), celiac disease, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
14. Patients with an active non-infectious pneumonitis
15. History of primary immunodeficiency
16. History of allogeneic organ transplant
17. Known history of previous clinical diagnosis of tuberculosis
18. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab. Inactivated viruses, such as those in the influenza vaccine, are permitted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 785 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Patient Overall survival (OS) | from randomisation until date of death from any cause (follow-up until 8 years post-treatment)
  defined as the interval in whole days between date of randomisation and date of death from any cause
Patient Event Free Survival (EFS) | From randomisation until date of progression/persistence/recurrence/death (follow-up until 8 years post-treatment)
  defined as the interval in whole days between date of randomisation until date of progression/persistence/recurrence/death

SECONDARY OUTCOMES:
Number of Acute (<3 months post-treatment) toxicity events experienced | From date of randomisation until 2 year follow-up
  Total number of acute (<3 months post-treatment) severe (grade 3-5) toxicity events experienced. Adverse events will be collected post-treatment and graded according to Common Terminology Criteria for Adverse Events (CTCAE).
Number of late (up to 2 years post-treatment) toxicity events experienced using CTCAE | From date of randomisation until 2 year follow-up
  Severe (grade 3-5) adverse events will be collected up to 2 years post randomisation, these events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and version 3.0 for scoring mucositis.
Number of late (up to 2 years post-treatment) toxicity events experienced using RTOG | From date of randomisation until 2 year follow-up
  Late and severe toxicity events at 2 years post randomisation,will be collected and graded using Radiation Therapy Oncology Group (RTOG) Radiation Morbidity Scoring Criteria
Head and neck specific quality of life at 2 years post-randomisation using EORTC C30 | From date of randomisation until 2 year follow-up
  Patients will complete the European Organisation for Research and Treatment of Cancer (EORTC) C30 questionnaire at baseline, at the end of treatment, and during the follow-up period until 2 years post-treatment
Head and neck specific Quality of Life at 2 years post-randomisation | From date of randomisation until 2 year follow-up
  Patients will complete the European Organisation for Research and Treatment of Cancer (EORTC) H&N35 questionnaire at baseline, at the end of treatment, and during the follow-up period until 2 years post-treatment
Swallowing outcomes assessed using MDADI Questionnaire at 24 months post-chemoradiotherapy | From date of randomisation until 2 year follow-up
  Patients will complete the M.D. Anderson Dysphagia Inventory (MDADI) Questionnaire at baseline, at the end of treatment, and during the follow-up period until 2 years post-treatment
Levels of Percutaneous Endoscopic Gastrostomy (PEG) use | From date of randomisation until 2 year follow-up
  PEG use will be assessed at baseline, throughout treatment and during 2 year follow-up period
Cost effectiveness of treatment as assessed using EuroQol Group (EQ-5D) questionnaire | From date of randomisation until 2 year follow-up
  Patients will complete the EuroQol Group (EQ-5D) questionnaire at baseline, at the end of treatment, and during the follow-up period until 2 years post-treatment
Surgical complication rates in each arm for patients who require a neck dissection at 4 months following the 3 month post-chemoradiotherapy assessment scan. | At 4 months following the 3 month post-chemoradiotherapy scan
  Surgical complication rates will be assessed at trial visits if a neck dissection is required at 4 months post-chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Prof Mehanna, Principal Investigator — University of Birmingham
Locations (38):
- Ireland (2):
  - St Luke's Hospital, Dublin
  - St James's Hospital, Dublin
- United Kingdom (36):
  - Royal Devon and Exeter Hospital, Exeter, Devon
  - Leicester Royal Infirmary, Leicester, East Midlands
  - Castle Hill Hospital, Cottingham, East Yorkshire
  - Colchester General Hospital, Colchester, Essex
  - Queen's Hospital, Romford, Essex
  - Royal Preston Hospital, Preston, Lancashire
  - James Cook University Hospital, Middlesbrough, North Yorkshire
  - York Hospital, York, North Yorkshire
  - Churchill Hospital, Oxford, Oxfordshire
  - Weston Park Hospital, Sheffield, South Yorkshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - University Hospital Coventry, Coventry, West Midlands
  - Newcross Hospital, Wolverhampton, West Midlands
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - St James's University Hospital, Leeds, West Yorkshire
  - Aberdeen Royal Infirmary, Aberdeen
  - Royal United Hospital, Bath
  - Belfast City Hospital, Belfast
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Aintree University Hospital, Liverpool
  - North Middlesex Hospital, London
  - Christie Hospital, Manchester
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Norfolk and Norwich University Hospital, Norwich
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - Royal Shrewsbury Hospital, Shrewsbury
  - Singleton Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: No